CLINICAL TRIAL: NCT00001077
Title: An Open-Label, Randomized, Three-Arm, Comparative Trial of a Caloric Supplement With Peptides and Medium-Chain Triglycerides Versus a Caloric Supplement With Whole Protein and Long-Chain Triglycerides Versus No Caloric Supplement for the Prevention of Weight Loss in Individuals With AIDS Who Take a Daily Multivitamin and Mineral Supplement
Brief Title: A Comparison of Two Caloric Supplements in the Prevention of Weight Loss in Patients With AIDS Who Take Daily Multivitamin and Mineral Supplements
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: CPCRA 038; 11588 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: HIV Infections; HIV Wasting Syndrome
Keywords: Weight Loss; Acquired Immunodeficiency Syndrome; Nutritional Support
MeSH Terms: conditions — HIV Infections; HIV Wasting Syndrome; Weight Loss; Acquired Immunodeficiency Syndrome | interventions — Geritol; Peptamen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collection

GROUPS / COHORTS (3):
- 1: Participants will receive peptamen drinks and multivitamin and mineral supplements, taken in addition to a regular diet for 4 months
  Interventions: Dietary Supplement: Multivitamin and mineral supplements; Dietary Supplement: Peptamen
- 2: Participants will receive NuBasics drinks or equivalent amounts of NuBasics soups or bars and daily multivitamin and mineral supplements, taken in addition to a regular diet for 4 months
  Interventions: Dietary Supplement: Multivitamin and mineral supplements; Dietary Supplement: NuBasics
- 3: Participants will receive multivitamin and mineral supplements, taken in addition to a regular diet for 4 months
  Interventions: Dietary Supplement: Multivitamin and mineral supplements

INTERVENTIONS:
Dietary Supplement: Multivitamin and mineral supplements — Oral tablets taken daily
Dietary Supplement: Peptamen — Solution received daily
  Groups: 1
Dietary Supplement: NuBasics — Solution or dietary bar received daily
  Groups: 2

SUMMARY:
To compare a caloric supplement containing peptides and medium-chain triglycerides, a caloric supplement containing whole protein and long-chain triglycerides, and no caloric supplement for the prevention of weight loss in individuals with AIDS who take a daily multivitamin and mineral supplement.

DETAILED DESCRIPTION:
Patients will be randomized to one of 3 study arms:

Arm 1 - Peptamen drinks + multivitamin and mineral supplement, taken in addition to regular diet for 4 months Arm 2 - NuBasics drinks or equivalent amounts of NuBasics soups or bars + multivitamin and mineral supplement, taken in addition to regular diet for 4 months Arm 3 - Multivitamin and mineral supplement, taken in addition to regular diet for 4 months.

At months 0, 2, and 4, patients will be assessed for weight, body cell mass, patient-reported physical activity level, and dietary intake (by 24-hour dietary recall). At months 2 and 4, they will also be assessed for compliance with study regimen. Patients who complete their 4 month follow up visit will be provided with a 30 day supply of the caloric supplement of their choice (Peptamen or NuBasics) and a 30 day supply of the study multivitamin supplement.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* Stable weight.
* CD4+ cell count <200 cells/mm3.
* Life expectancy of at least 6 months.
* Parent or legal guardian to sign written, informed consent for patients < 18 years old.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* Active opportunistic infection, requiring acute treatment.
* Malignancy (other than stable cutaneous Kaposi's sarcoma that does not require systemic chemotherapy).
* Diabetes mellitus or other conditions requiring special dietary restrictions.
* Body mass index (BMI) >= 29.0 kg/m2.
* Disorders or conditions that, in the treating clinician's opinion, may prevent adequate compliance with protocol requirements.

Concurrent Medication:

Excluded:

* Growth hormone.
* Megestrol acetate (Megace).
* Cyproheptadine (Periactin).
* Dronabinol (Marinol).
* Thalidomide.
* Anabolic steroids (e.g., nandrolone decanoate)(Deca-durabolin).
* Pharmacologic-dose corticosteroids (e.g., > 15 mg/day prednisone equivalent)

NOTE:

* Men requiring testosterone replacement therapy for documented hypogonadism may be enrolled.
* Caloric nutritional supplements deemed by the clinician to promote weight gain or maintenance.

Patients with the following prior condition are excluded:

* History of phenylketonuria.

Prior Medication:

Excluded within the past 2 weeks:

* Use of caloric nutritional supplements for more than 5 days deemed by the clinician to promote weight gain or maintenance.

Excluded within the past 30 days:

* Growth hormone.
* Megestrol acetate (Megace).
* Cyproheptadine (Periactin).
* Dronabinol (Marinol).
* Thalidomide.
* Anabolic steroids (e.g., nandrolone decanoate)(Deca-durabolin)
* Pharmacologic-dose corticosteroids (e.g., > 15 mg/day prednisone equivalent).

NOTE:

* Men requiring testosterone replacement therapy for documented hypogonadism may be enrolled.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV-infected participants who take a daily multivitamin and mineral supplement
Sampling Method: Non-Probability Sample
Enrollment: 536 (Actual)
Dates: Start 1996-06; Primary Completion 1998-04 (Actual); Study Completion 1998-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert CL, Study Chair; Wheeler D, Study Chair
Locations (17):
- United States (17):
  - Community Consortium / UCSF, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Washington Reg AIDS Prog / Dept of Infect Dis, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Baltimore Trials, Baltimore, Maryland
  - Wayne State Univ / WSU / DMC HIV / AIDS Program, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Southern New Jersey AIDS Cln Trials / Dept of Med, Camden, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Partners in Research - New Mexico, Albuquerque, New Mexico
  - Partners Research, Albuquerque, New Mexico
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Gibert CL, Muurahainen N, Collins G, Williams B, Raghavan S, Bartsch G, Wheeler D. Body composition in HIV-infected men and women in 1996-1997 (CPCRA 038). Int Conf AIDS. 1998;12:554 (abstract no 32169)
- [Background] Williams SB, Collins G, Muurahainen N, Bartsch G, Gibert C, Raghavan SS, Wheeler D. Protein intake is associated with body cell mass in weight-stable HIV+ men with CD4 < 200 cells/mm3: CPCRA 038. Int Conf AIDS. 1998;12:841-2 (abstract no 42339)
- [Background] Muurahainen N, Mulligan K. Clinical trials update in human immunodeficiency virus wasting. Semin Oncol. 1998 Apr;25(2 Suppl 6):104-11. PMID 9625392
- [Background] Muurahainen N, Collins G, Wheeler D, Mateo N, Madans M, Bartsch G, Gilbert C. Body cell mass (BCM) in HIV-infected (HIV+) males in the community programs for clinical research on AIDS (CPCRA) in 1996-1997. Int Conf AIDS. 1998;12:840 (abstract no 42333)
- [Background] Gibert CL, Wheeler DA, Collins G, Madans M, Muurahainen N, Raghavan SS, Bartsch G. Randomized, controlled trial of caloric supplements in HIV infection. Terry Beirn Community Programs for Clinical Research on AIDS. J Acquir Immune Defic Syndr. 1999 Nov 1;22(3):253-9. doi: 10.1097/00126334-199911010-00006. PMID 10770345